CLINICAL TRIAL: NCT06093841
Title: Relmacabtagene Autoleucel As Second-Line Therapy in Adult Patients with Aggressive B-cell NHL: a Single-arm, Multicenter, Open, Phase II Study
Brief Title: Relmacabtagene Autoleucel As Second-Line Therapy in Adult Patients with Aggressive B-cell NHL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029216
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Follicular Lymphoma Grade 3B; High-grade B-cell Lymphoma; Mediastinal B-Cell Diffuse Large Cell Lymphoma
Keywords: Relmacabtagene Autoleucel; aggressive B-cell non-Hodgkin lymphoma; Chimeric antigen receptor T cells; second-line
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — relmacabtagene autoleucel; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Relmacabtagene Autoleucel (Experimental): Experimental: Relmacabtagene Autoleucel Participants will receive cyclophosphamide250 mg/m^2/day intravenously (IV) and fludarabine 25 mg/m^2/day IV conditioning chemotherapy for 3 days followed by Relmacabtagene Autoleucel administered as a single IV infusion at a target dose of 1 x 10^8 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells on Day1.
  Interventions: Biological: Relmacabtagene Autoleucel; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Relmacabtagene Autoleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: JWCAR029
Drug: Fludarabine — Administered according to package insert
Drug: Cyclophosphamide — Administered according to package insert

SUMMARY:
The primary objective of this study is to asess the efficacy of Relmacabtagene autoleucel as second-line therapy in adult patients with aggressive B-cell Non-Hodgkins Lymphoma who are ineligible for haematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 2 study to determine the antitumor activity, PK, and safety of JWCAR029(Relmacabtagene autoleucel ) in subjects who have relapsed within 12 months from, or are refractory to, a single line of immunochemotherapy for aggressive Bcell NHL and are ineligible for HSCT (as defined in the eligibility criteria). Subjects will be treated with lymphodepleting chemotherapy and JWCAR029.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. Signed written informed consent obtained prior to any study procedures;
3. Histologically confirmed relapsed or refractory (R/R) aggressive B-cell NHL of the following histologiesLBCL as defined by the World Health Organization (WHO) Classification 2022:Diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS), high-grade B-cell lymphoma (HGL) with MYC and BCL2 rearrangements,HGL-NOS, Primary mediastinal large B-cell lymphoma, Follicular lymphoma Grade 3B (FL3B),Indolent B-NHL-transformed large B-cell lymphoma with adequate prior treatment with anthracycline-containing agents and rituximab or other CD20-targeted agents;
4. Subjects must meet the definition of refractory or relapsed;
5. Subjects were not eligible for HDCT/ASCT based on the investigator's assessment ;
6. Adequate organ function;
7. Presence of positive PET assessable lesions as determined by the Lugano criteria ;
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
9. Expected survival greater than 12 weeks;
10. Adequate vascular access for leukapheresis procedure;
11. Women of childbearing potential must agree to use highly effective methods of contraception for at least 28 days prior to lymphocyte clearance chemotherapy through 2 year after Relmacabtagene Autoleucel infusion; Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 2 year after Relmacabtagene Autoleucel infusion;

Exclusion Criteria:

1. Subjects with non-Hodgkin's lymphoma who have received second or more line therapy;
2. Lymphoma of the primary center (subjects with secondary central nervous system lymphoma are allowed to enroll;
3. History of another primary malignancy that has not been in remission for at least 2 years;
4. Subjects has active HBV, HCV, HIV or syphilis infection at the time of screening;
5. Deep venous thrombosis (DVT)/Pulmonary embolism (PE), or DVT/PE requires anti-coagulation within 3 months prior to signing the ICF;
6. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection;
7. Uncontrolled diabetes and hypertension;
8. Presence of acute or chronic graft-versus-host disease (GVHD);
9. Active autoimmune disease requiring immunosuppressive therapy;
10. History of any serious cardiovascular disease or presence of clinically relevant CNS pathology;
11. Pregnant or nursing women;
12. Subjects Received an autologous or allogeneic hematopoietic stem cell transplant;
13. Uncontrolled conditions or unwillingness or inability to follow the procedures required in the protocol;
14. Received CAR T-cell or other genetically-modified T-cell therapy previously;
15. Received live vaccination within 6 weeks prior to lymphocyte clearance chemotherapy;
16. History of severe hypersensitivity reactions to any of the drug ingredients used in this study product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2029-11-04 (Estimated)

PRIMARY OUTCOMES:
ORR at 3 month | 3 months
  Percentage of participants with CR [CMR;CRR] or PR [partial metabolic response (PMR);

SECONDARY OUTCOMES:
CRR at 3 month | 3 months
  Complete response rate in subjects at 3 month
Duration of response (DOR) | up to 2 years after Relmacabtagene Autoleucel infusion
  Time from first response(PR or CR) to disease progression or death from any cause.
Duration of complete remission (DoCR) | up to 2 years after Relmacabtagene Autoleucel infusion
  Time from complete response (CR) to disease progression or death from any cause.
Duration of partial remission (DoPR) | up to 2 years after Relmacabtagene Autoleucel infusion
  Time from partial response (PR) to disease progression or death from any cause.
Time to response (TTR) | up to 2 years after Relmacabtagene Autoleucel infusion
  Time from JWCAR029 infusion to first documentation of CR or PR
Progression-Free Survival (PFS) | up to 2 years after Relmacabtagene Autoleucel infusion
  PFS is defined as the time from the Relmacabtagene Autoleucel infusion date to the date of disease progression per Lugano classification or death from any cause.
Overall Survival (OS) | up to 2 year after Relmacabtagene Autoleucel infusion
  OS is defined as the time from Relmacabtagene Autoleucel infusion to the date of death from any cause.
Adverse events (AEs) | up to 2 year after Relmacabtagene Autoleucel infusion
  Types, frequency, and severity of adverse events and laboratory anomalies Physiological parameter
Pharmacokinetic (PK)- Cmax of Relmacabtagene Autoleucel | up to 1 year after Relmacabtagene Autoleucel infusion
  Maximum observed concentration of Relmacabtagene Autoleucel in peripheral blood
Pharmacokinetic (PK)- Tmax of Relmacabtagene Autoleucel | up to 1 year after Relmacabtagene Autoleucel infusion
  Time to maximum concentration of Relmacabtagene Autoleucel in peripheral blood
Pharmacokinetic (PK)- AUC of Relmacabtagene Autoleucel | up to 1 year after Relmacabtagene Autoleucel infusion
  Area under the concentration vs time curve of Relmacabtagene Autoleucel
The concentration of Car-T cell | up to 1 year after Relmacabtagene Autoleucel infusion
  The concentration of Car-T cell in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, PhD, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Depei Wu, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (13):
- China (13):
  - Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine,, Shanghai, Shanghai Municipality
  - Institute of Hematology&Hospital of Blood Disease CAMS, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Jiangsu Provincial People's Hospital, Nanjing

IPD SHARING:
Plan to Share IPD: No